CLINICAL TRIAL: NCT03947684
Title: EMRSHN 2: Exploring the Modulatory Role of Sex Hormones Along the Neuromechanical Axis in Females
Brief Title: Exploring the Modulatory Role of Sex Hormones Along the Neuromechanical Axis in Females
Acronym: EMRSHN
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Yasin Dhaher, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2018-0192; 1R01AR069176-01A1 (NIH)
Record Dates: First submitted 2019-04-22; First posted 2019-05-13 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Role of Sex Hormones Along the Neuromechanical Axis
Keywords: Sex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected every other day for a period of two months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Non-Oral Contraceptive (NOC): Females ages 18-39 years, who are eumenorrheic (regular monthly cycles of 24-35 days) and moderately active. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, pacemaker, metal implants in the head region, history of epilepsy or seizures, skull fractures or skull deficits, concussion within the last 6 months, unexplained recurring headaches, medications that lower seizure threshold, and pregnancy.
- Oral Contraceptive ( OC): Females: ages 18-39 years, who are on a stable hormonal contraceptive regimen for 6 months (oral, transdermal or vaginal) and moderately active. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, started or stopped taking oral contraceptives within the previous 6 months, participate in high impact endurance training (i.e. pre-marathon training, body building), or currently participating in competitive level sports.
- Male: Males: Ages 18-39. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, pacemaker, metal implants in the head region, history of epilepsy or seizures, skull fractures or skull deficits, concussion within the last 6 months, unexplained recurring headaches, and medications that lower seizure threshold.

SUMMARY:
The goal of this project is to test our central hypothesis that changes in sex hormone concentration result in changes to the basic elements of motor control - at multiple levels, from the musculotendinous unit to motor control circuitry. Under Aim 1 the investigator will determine the influence of sex hormone fluctuations on the muscle stretch reflex during active and passive states, and the time lag between hormone concentration changes and the reflex response. The investigator will use a technically simple assessment that could be implemented in the field. Under Aim 2 the investigator will determine the influence of sex hormone fluctuations on spinal motor neuron excitability using H-reflex as a probe and the simultaneous change in the muscle mechanics using muscle twitch response. Aims 1 & 2 will include a focus on the differential role of oral contraceptives. In Aim 3 the investigator will use paired-pulse transcranial magnetic stimulation during active contraction to determine the influence of sex hormone fluctuation.

ELIGIBILITY:
Inclusion Criteria:

* Females: ages 18-39 years, who are eumenorrheic (regular monthly cycles of 24-35 days) or on a stable hormonal contraceptive regimen for 6 months (oral, transdermal or vaginal), no history of pregnancy, moderately active (less than 7 hours of vigorous physical activity per week)
* Males: Ages 18-39

Exclusion Criteria:

* History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, current smoker, history of disordered eating, history of stress fracture in the lower limb, history of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease).
* For female participants only: Point of care screening for anemia will be completed, and individuals with hemoglobin levels <11.6 g/dl will be excluded from participating in the study.
* Specific exclusion criteria for TMS (male and female): pacemaker, metal implants in the head region, history of epilepsy or seizures, skull fractures or skull deficits, concussion within the last 6 months, unexplained recurring headaches, medications that lower seizure threshold, and pregnancy.
* Additional exclusion criteria for female participants: History of menstrual dysfunction (primary or secondary amenorrhea, oligomenorrhea, anovulatory cycles, polycystic ovarian disease), current or past pregnancy, started or stopped taking oral contraceptives within the previous 6 months, exercise vigorously more than 7 hours per week or currently participating in competitive level sports. The reason for excluding highly active or competitive athletes is due to the high rate of undiagnosed menstrual dysfunction in females of this population.
* This study will not include: adults unable to consent, Individuals who are not yet adults (infants, children, teenagers), pregnant women or prisoners.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Non oral contraceptive group (NOC): Healthy females at 18-39 years old, who are eumenorrheic (regular monthly cycles of 24-35 days) and moderately active;
  Oral contraceptive group (OC): Healthy females at 18-39 years old, who are on a stable hormonal contraceptive regimen for 6 months (oral, transdermal or vaginal) and moderately active;
  Male group: Healthy males at 18-39 years old.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasin Dhaher, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Oral Contraceptive (NOC): Females: ages 18-39 years, who are eumenorrheic (regular monthly cycles of 24-35 days) and moderately active. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, history of menstrual dysfunction (primary or secondary amenorrhea, oligomenorrhea, anovulatory cycles, polycystic ovarian disease), current pregnancy, started or stopped taking oral contraceptives within the previous 6 months, participate in high impact endurance training (i.e. pre-marathon training, body building), or currently participating in competitive level sports. Specific exclusion criteria for TMS: pacemaker, metal implants in the head region, history of epilepsy or seizures, skull fractures or skull deficits, concussion within the last 6 months, unexplained recurring headaches, medications that lower seizure threshold.
- Oral Contraceptive (OC): Females: ages 18-39 years, who are on a stable hormonal contraceptive regimen for 6 months (oral, transdermal or vaginal) and moderately active. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, started or stopped taking oral contraceptives within the previous 6 months, participate in high impact endurance training (i.e. pre-marathon training, body building), or currently participating in competitive level sports.
- Male: Ages 18-39. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, pacemaker, metal implants in the head region, history of epilepsy or seizures, skull fractures or skull deficits, concussion within the last 6 months, unexplained recurring headaches, medications that lower seizure threshold.
Period: Overall Study
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Started | 61 | 30 | 11
Completed | 34 | 21 | 10
Not Completed | 27 | 9 | 1
Not completed — Lost to Follow-up | 13 | 5 | 1
Not completed — Withdrawal by Subject | 11 | 4 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lack of adherence to study protocol | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Oral Contraceptive (NOC): Females: ages 18-39 years, who are eumenorrheic (regular monthly cycles of 24-35 days) and moderately active. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, history of menstrual dysfunction (primary or secondary amenorrhea, oligomenorrhea, anovulatory cycles, polycystic ovarian disease), current pregnancy, started or stopped taking oral contraceptives within the previous 6 months, participate in high impact endurance training, or currently participating in competitive level sports. Specific exclusion criteria for TMS: pacemaker, metal implants in the head region, history of epilepsy or seizures, skull fractures or skull deficits, concussion within the last 6 months, unexplained recurring headaches, medications that lower seizure threshold, and pregnancy.
- Oral Contraceptive (OC): Females: ages 18-39 years, who are on a stable hormonal contraceptive regimen for 6 months (oral, transdermal or vaginal) and moderately active. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, started or stopped taking oral contraceptives within the previous 6 months, participate in high impact endurance training, or currently participating in competitive level sports.
- Total: Total of all reporting groups
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male | Total
Number analyzed (Participants) | 61 | 30 | 11 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 61 | 30 | 11 | 102
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (5) | 27 (4) | 28 (5) | 27 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 30 | 0 | 91
  Male | 0 | 0 | 11 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 5 | 0 | 18
  Not Hispanic or Latino | 36 | 21 | 11 | 68
  Unknown or Not Reported | 12 | 4 | 0 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 5 | 8 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 1 | 8
  White | 32 | 19 | 2 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 4 | 0 | 17
Region of Enrollment [Number; unit: participants]
  United States | 61 | 30 | 11 | 102

OUTCOME MEASURES:

1. Primary Outcome: Changes in Short-interval Intracortical Inhibition (SICI) During the Follicular Phase
Description: The conditioned motor evoked potential (MEP) at each inter-stimulus interval (ISI) was normalized to MEP obtained from unconditioned stimulation. Change was evaluated by regressing the normalized conditioned motor evoked potential amplitude at each ISI with estradiol concentration. Average and standard deviation for each ISI reported.
Time Frame: day 1 menses up to day with highest estradiol concentration
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: ratio to the unconditioned stimulus MEP
Groups:
- Non-Oral Contraceptive (NOC): Females ages 18-39 years, who are eumenorrheic (regular monthly cycles of 24-35 days) or on a stable hormonal contraceptive regimen for 6 months (oral, transdermal or vaginal) and moderately active. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, pacemaker, metal implants in the head region, history of epilepsy or seizures, skull fractures or skull deficits, concussion within the last 6 months, unexplained recurring headaches, medications that lower seizure threshold, and pregnancy.
  Additional exclusion criteria for female participants: History of menstrual dysfunction (primary or secondary amenorrhea, oligomenorrhea, anovulatory cycles, polycystic ovarian disease), current pregnancy, started or stopped taking oral contraceptives within the previous 6 months, participate in high impact endurance training (i.e. pre-marathon training, body building), or currently participating in competitive level sports.
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 17 | 0 | 0
ratio to the unconditioned stimulus MEP
  2 ms | 0.78 (0.21) |  |
  3 ms | 0.83 (0.22) |  |
  4 ms | 0.93 (0.24) |  |
  5 ms | 1.03 (0.26) |  |
  6 ms | 1.08 (0.37) |  |
  7 ms | 1.11 (0.20) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05; Test type: Other — Generalized linear model (GLM) with log link function and exchangeable correlation structure; p > 0.05, F-test

2. Primary Outcome: Change in Stretch Reflex at Relaxed State
Description: Muscle stretch reflex (MSR) was calculated by dividing the root mean squared (RMS) value of the electromyogram (EMG) response with the RMS of the muscle's EMG during maximal voluntary contraction and the force of the tapper used to elicit the reflex. Change was evaluated by regressing the ratio simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. Average and standard deviation for each menstrual phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: ratio to RMS MVC and tapper force
Groups:
- Non-Oral Contraceptive (NOC): Females: ages 18-39 years, who are eumenorrheic (regular monthly cycles of 24-35 days) and moderately active. Exclusion criteria: History of musculoskeletal or orthopedic injury of the spine, hip, knee, ankle or foot, history of neurological injury of the peripheral or central nervous system, history of disordered eating, of a connective tissue disorder (Marfan's syndrome, Ehlers-Danlos disease), history of or current diabetes, history of menstrual dysfunction (primary or secondary amenorrhea, oligomenorrhea, anovulatory cycles, polycystic ovarian disease), current pregnancy, started or stopped taking oral contraceptives within the previous 6 months, participate in high impact endurance training (i.e. pre-marathon training, body building), or currently participating in competitive level sports.
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 13 | 0 | 0
ratio to RMS MVC and tapper force
  Follicular | 0.0164 (0.0144) |  |
  Luteal | 0.0138 (0.0136) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test

3. Primary Outcome: Change in Spinal Motor Neuron Excitability in Non Oral Contraceptive User
Description: The spinal motor neuron excitability was measured by calculating the ratio between the maximum peak-to-peak value of H reflex and the maximum peak-to-peak value of M wave. Change was evaluated by regressing the ratio simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. Average and standard deviation for each menstrual phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: ratio to the max peak-to-peak M wave
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 24 | 0 | 0
ratio to the max peak-to-peak M wave
  Follicular | 0.6 (0.24) |  |
  Luteal | 0.61 (0.25) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

4. Primary Outcome: Normalized Conditioned Motor Evoked Potential in Male and Female
Description: The conditioned motor evoked potential (MEP) at each inter-stimulus interval (ISI) was normalized to MEP obtained from unconditioned stimulation. The difference between male and female groups was evaluated using a 2 (male vs. female) x 7 (ISI) repeated measures ANOVA. Average and standard deviation for each ISI reported.
Time Frame: menses period for female, day 1 for male
Population: Participants in NOC and male groups.
Measure: Mean (Standard Deviation); unit: ratio to the unconditioned stimulus MEP
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 17 | 0 | 10
ratio to the unconditioned stimulus MEP
  2 ms | 0.75 (0.22) |  | 1.02 (0.2)
  7 ms | 1.06 (0.2) |  | 1.17 (0.31)
  10 ms | 1.3 (0.35) |  | 1.35 (0.58)
  15 ms | 1.5 (0.51) |  | 1.24 (0.58)
  20 ms | 1.48 (0.71) |  | 1.22 (0.52)
  25 ms | 1.38 (0.74) |  | 1.16 (0.41)
  30 ms | 1.26 (0.74) |  | 0.99 (0.3)
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC) vs Male; Significance was accepted for p values <0.05; Test type: Other — Repeated measures ANOVA; p > 0.05, F-test

5. Primary Outcome: Change in Spinal Motor Neuron Excitability in Oral Contraceptive User
Description: The spinal motor neuron excitability was measured by calculating the ratio between the maximum peak-to-peak value of H reflex and the maximum peak-to-peak value of M wave. Change was evaluated by regressing the ratio simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. Average and standard deviation for active and inactive pill phase are reported.
Time Frame: Active pill, Inactive pill
Population: Participants in OC group.
Measure: Mean (Standard Deviation); unit: ratio to the max peak-to-peak M wave
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 0 | 17 | 0
ratio to the max peak-to-peak M wave
  Active pill |  | 0.67 (0.19) |
  Inactive pill |  | 0.67 (0.16) |
Statistical Analysis 1: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data obtained during active pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data obtained during inactive pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test

6. Secondary Outcome: Change in Steadiness of Isometric Force Production at 20% of Maximum Voluntary Contraction in Non Oral Contraceptive User
Description: Steadiness of the exerted force is quantified using coefficient of variation. Change was evaluated by regressing the steadiness simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) follicular phase, and (2) luteal phase. Average and standard deviation for each phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 7 | 0 | 0
percentage (%)
  Follicular | 2.2 (0.7) |  |
  Luteal | 2.2 (0.9) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test

7. Secondary Outcome: Change in Flexion Reflex Root Mean Squared Value in Non Oral Contraceptive User
Description: The root mean squared (RMS) value were calculated and averaged for each testing visit. Change was evaluated by regressing the RMS simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) follicular phase, and (2) luteal phase. Average and standard deviation for each phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: millivolt
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 24 | 0 | 0
millivolt
  Follicular | 0.093 (0.066) |  |
  Luteal | 0.111 (0.08) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

8. Secondary Outcome: Change in Flexion Reflex Duration in Non Oral Contraceptive User
Description: The duration were calculated and averaged for each testing visit. Change was evaluated by regressing the duration simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) follicular phase, and (2) luteal phase. Average and standard deviation for each phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 24 | 0 | 0
milliseconds
  Follicular | 36.58 (13.24) |  |
  Luteal | 35.60 (13.11) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

9. Secondary Outcome: Change in Flexion Reflex Latency in Non Oral Contraceptive User
Description: The latency measured from the onset of the stimulus were calculated and averaged for each testing visit. Change was evaluated by regressing the latency simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) follicular phase, and (2) luteal phase. Average and standard deviation for each phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 24 | 0 | 0
milliseconds
  Follicular | 81.96 (7.17) |  |
  Luteal | 80.73 (7.63) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test

10. Secondary Outcome: Change in Flexion Reflex Root Mean Squared Value in Oral Contraceptive User
Description: The root mean squared (RMS) value were calculated and averaged for each testing visit. Change was evaluated by regressing the RMS simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) active pill, and (2) inactive pill. Average and standard deviation for each phase is reported.
Time Frame: Active pill, Inactive pill
Population: Participants in OC group.
Measure: Mean (Standard Deviation); unit: millivolt
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 0 | 18 | 0
millivolt
  Active pill |  | 0.107 (0.074) |
  Inactive pill |  | 0.083 (0.034) |
Statistical Analysis 1: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during active pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during inactive pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

11. Secondary Outcome: Change in Flexion Reflex Duration in Oral Contraceptive User
Description: The duration were calculated and averaged for each testing visit. Change was evaluated by regressing the duration simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) active pill, and (2) inactive pill. Average and standard deviation for each phase is reported.
Time Frame: Active pill, Inactive pill
Population: Participants in OC group.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 0 | 18 | 0
milliseconds
  Active pill |  | 30 (5.71) |
  Inactive pill |  | 28.2 (6.23) |
Statistical Analysis 1: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during active pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during inactive pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test

12. Secondary Outcome: Change in Flexion Reflex Latency in Oral Contraceptive User
Description: The latency measured from the onset of the stimulus were calculated and averaged for each testing visit. Change was evaluated by regressing the latency simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) active pill, and (2) inactive pill. Average and standard deviation for each phase is reported.
Time Frame: Active pill, Inactive pill
Population: Participants in OC group.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 0 | 18 | 0
milliseconds
  Active pill |  | 77.7 (5.59) |
  Inactive pill |  | 76.4 (6.98) |
Statistical Analysis 1: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during active pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test
Statistical Analysis 2: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during inactive pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test

13. Other Pre Specified Outcome: Change in Muscle Twitch Peak Torque in Non Oral Contraceptive User
Description: Change was evaluated by regressing the peak torque simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) follicular phase, and (2) luteal phase. Average and standard deviation for each phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 20 | 0 | 0
Nm
  Follicular | 12.7 (2.49) |  |
  Luteal | 12.4 (2.44) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained from follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained from luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

14. Other Pre Specified Outcome: Number of Positive Ovulation
Description: Urinary ovulation kits is used to verify the ovulatory cycles and identify the approximate day of ovulation of the NOC group.
Time Frame: Follicular
Population: Participants in NOC group.
Measure: Number; unit: positive ovulation
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 61 | 0 | 0
positive ovulation | 53 |  |

15. Other Pre Specified Outcome: Change in Muscle Twitch Time to Peak Torque in Non Oral Contraceptive User
Description: Change was evaluated by regressing the time to peak torque simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) follicular phase, and (2) luteal phase. Average and standard deviation for each phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 20 | 0 | 0
milliseconds
  Follicular | 94.6 (14) |  |
  Luteal | 91 (12.1) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained from follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained from luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

16. Other Pre Specified Outcome: Change in Muscle Twitch Half Relaxation Time in Non Oral Contraceptive User
Description: Change was evaluated by regressing the half relaxation time simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) follicular phase, and (2) luteal phase. Average and standard deviation for each phase is reported.
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 20 | 0 | 0
milliseconds
  Follicular | 119 (21.3) |  |
  Luteal | 115 (20) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained from follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained from luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test

17. Other Pre Specified Outcome: Change in Muscle Twitch Peak Torque in Oral Contraceptive User
Description: Change was evaluated by regressing the peak torque simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) active pill, and (2) inactive pill. Average and standard deviation for each phase is reported.
Time Frame: Active pill, Inactive pill
Population: Participants in OC group.
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 0 | 18 | 0
Nm
  Active pill |  | 13.9 (5.06) |
  Inactive pill |  | 14.3 (5.96) |
Statistical Analysis 1: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during active pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during inactive pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

18. Other Pre Specified Outcome: Change in Muscle Twitch Time to Peak Torque in Oral Contraceptive User
Description: Change was evaluated by regressing the time to peak torque simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) active pill, and (2) inactive pill. Average and standard deviation for each phase is reported.
Time Frame: Active pill, Inactive pill
Population: Participants in OC group.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 0 | 18 | 0
milliseconds
  Active pill |  | 98.1 (19.2) |
  Inactive pill |  | 95 (14.4) |
Statistical Analysis 1: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during active pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test
Statistical Analysis 2: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during inactive pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

19. Other Pre Specified Outcome: Change in Muscle Twitch Half Relaxation Time in Oral Contraceptive User
Description: Change was evaluated by regressing the half relaxation time simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) active pill, and (2) inactive pill. Average and standard deviation for each phase is reported.
Time Frame: Active pill, Inactive pill
Population: Participants in OC group.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 0 | 18 | 0
milliseconds
  Active pill |  | 124 (21.5) |
  Inactive pill |  | 128 (18) |
Statistical Analysis 1: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during active pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test
Statistical Analysis 2: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during inactive pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

20. Secondary Outcome: Change in Steadiness of Isometric Force Production at 20% of Maximum Voluntary Contraction in Oral Contraceptive User
Description: Steadiness of the exerted force is quantified using coefficient of variation. Change was evaluated by regressing the steadiness simultaneously on estradiol and progesterone concentrations, and estradiol x progesterone interaction. The analyses was performed during (1) active pill, and (2) inactive pill. Average and standard deviation for each phase is reported.
Time Frame: Active pill, Inactive pill
Population: Participants in OC group.
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 0 | 7 | 0
percentage (%)
  Active pill |  | 1.9 (0.8) |
  Inactive pill |  | 1.9 (0.7) |
Statistical Analysis 1: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during active pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p < 0.05, Wald test
Statistical Analysis 2: Comparison: Oral Contraceptive (OC); Significance was accepted for p values <0.05. Data is obtained during inactive pill phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

21. Primary Outcome: Changes in Intracortical Facilitation (ICF) During the Follicular Phase
Description: as for outcome 1
Time Frame: day 1 menses up to day with highest estradiol concentration
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: ratio to the unconditioned stimulus MEP
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 17 | 0 | 0
ratio to the unconditioned stimulus MEP
  10 ms | 1.32 (0.38) |  |
  15 ms | 1.54 (0.51) |  |
  20 ms | 1.46 (0.59) |  |
  25 ms | 1.37 (0.62) |  |
  30 ms | 1.28 (0.64) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05; Test type: Other — Generalized linear model (GLM) with log link function and exchangeable correlation structure; p > 0.05, F-test

22. Primary Outcome: Change in Stretch Reflex at Active State
Description: as for outcome 2
Time Frame: Follicular, Luteal
Population: Participants in NOC group.
Measure: Mean (Standard Deviation); unit: ratio to RMS MVC and tapper force
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
Number analyzed (Participants) | 17 | 0 | 0
ratio to RMS MVC and tapper force
  Follicular | 0.0106 (0.00876) |  |
  Luteal | 0.0111 (0.0114) |  |
Statistical Analysis 1: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during follicular phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test
Statistical Analysis 2: Comparison: Non-Oral Contraceptive (NOC); Significance was accepted for p values <0.05. Data is obtained during luteal phase; Test type: Other — Generalized estimating equation (GEE) with log link function and exchangeable correlation structure; p > 0.05, Wald test

ADVERSE EVENTS:
Time Frame: Adverse event collection starts after the subject has provided informed consent, ends 30 days following the last research session, an average of 2 months for NOC group, 1 month for OC group, and 1 day for male group.
Arm/Group | Non-Oral Contraceptive (NOC) | Oral Contraceptive (OC) | Male
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/30 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/30 | 0/11
Other Adverse Events (participants affected / at risk) | 0/61 | 0/30 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT03947684/Prot_SAP_000.pdf